CLINICAL TRIAL: NCT02435446
Title: Comparison of Cone Beam With CT Scan for the Diagnosis of Otosclerosis
Brief Title: Cone Beam and CT Scan for the Diagnosis of Otosclerosis (TACOS)
Acronym: TACOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PROBLEM of inclusion
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MWS_2015_18
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Otosclerosis
MeSH Terms: conditions — Otosclerosis | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eligible patients for cone-beam (Experimental): A cone-beam computed tomography will be offered to the patients undergoing a CT scan for the diagnosis and/or the pre-operative assessment of an otosclerosis, fulfilling the inclusion criterias and without any exclusion criteria.
  Interventions: Device: Cone-beam computed tomography

INTERVENTIONS:
Device: Cone-beam computed tomography — Cone-beam computed tomography

SUMMARY:
Computed tomography scan (CT) is routinely used for the diagnosis and the pre-operative assessment of otosclerosis.

The cone-beam computed tomography (CBCT) is a imaging technique with reduced irradiating and, therefore, could replace the CT.

In this study, a CBCT will be proposed to all patients undergoing a CT exam for the diagnosis and/or the pre-operative assessment of an otosclerosis.

The results of the CBCT will be compared to those of the CT scan.

ELIGIBILITY:
Inclusion Criteria:

* CT scan indicated for the diagnosis and pre-operatice assessment of an otosclerosis

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Patient under a legal protection procedure
* Patient denying to participate to the study
* Lack of affiliation to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the cone-beam computed tomography vs CT scan assessed by the presence or absence of areas of sclerosis | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France